CLINICAL TRIAL: NCT05458050
Title: A Double-blind, Intervention, Post-marketing Investigation to Identify Subjects Who Are Admitted to Hospital With an Increased Risk of Developing Pressure Ulcers, Using PU Sensor
Brief Title: An Investigation to Identify Subjects Admitted to Hospital With an Increased Risk of Developing Pressure Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PU sensor AB (Industry)
Collaborators: Aurevia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CIP-PUS-1-001
Record Dates: First submitted 2022-06-15; First posted 2022-07-14 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: Double blind
Masking Description: The medical device will give an ID number but the results from the measurement will be masked until data base is locked (DBL). The data from the measurement will be available after DBL
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PU Sensor examination (Other): Device:PU Sensor will assess the microcirculation in sacrum with and without pressure (subject will lay on side and after that on back) the total measurement time is 5-10 minutes
  Interventions: Device: PU sensor

INTERVENTIONS:
Device: PU sensor — Device to assess microcirculation in sacrum area to find subjects at risk for pressure ulcer

SUMMARY:
A double blind, non randomized, multicenter investigation

DETAILED DESCRIPTION:
The study consists of 2 evaluations/visits.

Evaluation/visit 1: Takes place in connection with admission to the hospital. Informed consent, inclusion and exclusion criteria are assessed as well as assessment of skin type and inspection of the entire body skin. Pregnancy test on women of childbearing potential, height, weight, blood pressure and body temperature are measured. Questions about demography, health conditions, previous illnesses, nicotine habits. Risk assessment for pressure ulcers (Modified Norton or RAPS-scale) is carried out according to the hospital usual routine. Examination with PU sensor will be performed.

Evaluation/visit 2: Takes place in connection with the discharge from the hospital or 4 weeks after visit 1 if the research subject is still hospitalized. Full body skin inspection to see possible onset of pressure ulcers. Review of the research subject's medical records as well as review of nursing notes from the hospital where the research subject has been discharged from, to find any notes about pressure ulcers. The study participation is then terminated for the research subject.

ELIGIBILITY:
Inclusion Criteria:

1. Given their written consent to participate in the study
2. Male or female between ≥18 years and ≤ 64 years with a reduced mobility, where the hospitalization may involve a risk that the person may become less active or Male or female ≥65 years

Exclusion Criteria:

1. Existing pressure ulcer or damage to the skin around the sacrum where the PU sensor plate and pillow are to be placed
2. Fever ≥38 ºC, within 30 minutes before the examination with PU sensor
3. Difficulty lying still in supine position during the examination with PU sensor, which takes 5 to 10 minutes
4. Known allergy or sensitivity to any of the materials in PU sensor that gets in contact with the skin on the sacrum
5. Body weight ≥200 kg
6. Previous participation in the study
7. Mental inability, or language difficulties that results in difficulty to understand the meaning of participation in the study and / or signing the study consent,
8. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Number of pressure ulcers developed between visit 1 and 2 | Up to 4 weeks
  This outcome is to evaluate if the subjects that have been assessed as at risk of developing pressure ulcers (using PU sensor) have actually developed pressure ulcers with a greater probability than those assessed as not at risk

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) and adverse device effects (ADEs) | Up to 2 days
  All adverse events (AEs) and adverse device effects (ADEs) incidence and severity following measurement with PU sensor up to 2 days after the baseline

OTHER OUTCOMES:
Proportion of pressure ulcers located in sacrum | Up to 4 weeks
  The examination with PU sensor is in sacrum. Proportion of pressure ulcers that are located in sacrum for PU sensor high-risk group compared to PU sensor low-risk group.
  PU sensor high-risk group are those subjects who have a decreased blood flow at pressure from their own body, resulting in a "High risk" result from PU sensor.
  This proportion is compared for the two groups to evaluate if PU sensor can assess risk of pressure ulcers on the skin everywhere, or only in sacrum where the examination is done.
Combine Norton/RAPS with PU Sensor results | Up tp 4 weeks
  All subject will use Norton or RAPS for risk assessment of pressure ulcer. The results from these risk assessments will be compared with the results from PU Sensor and pressure ulcers developed to explore if a combination of the scales and PU sensor would give a better view of subjects at risk.
Compare PU sensor examinations for different skin types | Up to 4 weeks
  PU sensor is using PPG (Photoplethysmography) to assess blood flow in sacrum. Since light is used the the skin type (amount of pigment and in the skin etc) may affect the examination.
Compare PU sensor examinations for subjects with underlying disease | Up to 4 weeks
  PU sensor is using PPG (Photoplethysmography) to assess blood flow in sacrum. Underlying diseases such as Hypertension and/or Diabetes may affect the examination.

CONTACTS AND LOCATIONS:
Overall Officials: Anna-Christina Ek, RN,PhD, Study Chair — PU Sensor
Locations (3):
- Sweden (3):
  - Länssjukhuset Ryhov, Geriatriska kliniken, Jönköping
  - Oskarhamns Sjukhus, Oskarshamn
  - Medicin-Geriatriska kliniken Akademiska sjukhuset,, Uppsala

IPD SHARING:
Plan to Share IPD: No
Due to uncertainties in EU data protection legislation individual deidentified participant data are not shared. The main uncertainty is the concept of what "deidentified" means. It appears not to mean that the data set of a person is simply separated from the person's name. What additional operations have to be done appears to depend on technological capabilities to re-identify the persons associated with the data set. A common perception is that the technological capabilities for re-identification are permanently increasing. This could have the effect that public data sets that are regarded as deidentified now might become re-identifiable data sets in the future. Once this happens, the sponsor is no longer able to make the publication of the data sets un-happen. This could result in punishment by EU data protection authorities. The sponsor wants to avoid this.